CLINICAL TRIAL: NCT00197340
Title: Antepartum Chronic Epidural Therapy (ACET) Using Ropivacaine to Improve Uteroplacental Blood Flow in Pre-Eclampsia and Intrauterine Growth Restriction
Brief Title: Antepartum Chronic Epidural Therapy (ACET) to Improve Blood Flow to the Uterus, Placenta and Baby in Pre-Eclampsia and Intrauterine Growth Restriction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: International Anesthesia Research Society (IARS) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACET1-ginosar-HMO-CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2006-02

CONDITIONS: Pre-Eclampsia; Fetal Growth Retardation
Keywords: Pre-Eclampsia; Fetal Growth Retardation; Anesthesia, Epidural; Placental Circulation; Dose-Response Relationship, Drug
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

INTERVENTIONS:
Drug: Epidural ropivacaine

SUMMARY:
Pre-eclampsia (PE) and intrauterine growth restriction (IUGR) are common and important disorders of pregnancy. Both disorders are associated with an impairment of uteroplacental blood flow (UPBF). No effective therapy has been identified to reliably improve UPBF in these patients and typically, obstetric management involves interventional delivery, particularly problematic when remote from term. This study assess the hypothesis that epidural local anesthetics may improve UPBF in these patients.

DETAILED DESCRIPTION:
Women with sonographic uterine artery flow abnormalities and either PE or IUGR (or both) were randomized to either ACET or non ACET control. Both groups were able to receive standard therapies (in-hospital monitoring, magnesium and anti-hypertensives as appropriate). The first five days of the therapeutic arm (ACET) consisted of a dose-finding trial, where epidural ropivacaine infusions (10ml/hr for 24 hours) of 0•04%, 0•06%, 0•08% and 0•1% and a saline placebo were each administered via tunneled epidural catheters in a randomized, double-blinded, cross-over design over five consecutive days; all three women received all doses. Doppler measurement of flow in the uterine artery was performed at baseline and at the end of each dose period. The ideal dose for an individual was determined to be lowest dose of drug giving maximal effect without side effects; in the second stage of the study, this dose was administered until delivery with the addition of a second placebo day to during this period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Reliable gestational age based upon an ultrasound crown-rump length performed between 7 to 14 completed weeks gestation. If the ultrasound date matches the date of the last menstrual period (LMP) within 7 days, the LMP date is used, otherwise the ultrasound date is used.

  2. Gestational age at the time of enrollment between 28 to 32 weeks (based upon 1.) and need for in-hospital observation or treatment REGARDLESS of the study.

  3. Presence of uterine artery notching in ultrasound scan. 4. EITHER 4a or 4b (if both, the patient is enrolled as for 4a): 4a. Pre-eclampsia: Women must have criteria #1 and #2 Criterion #1: Hypertension (> 140/90) at rest, measured twice, at least 6 hours apart.

Criterion #2: Proteinuria:

EITHER: At least 0.1 g/l in two random samples at least 6 hours apart. OR: At least 0.3g in a 24 hour collection.

4b Intrauterine growth retardation (IUGR): Women must have criteria #1 and #2. Criterion #1: Ultrasound abdominal circumference below 10th percentile. Criterion #2: Established IUGR for at least 2 weeks.

Exclusion Criteria:

* at the time of enrollment: active labor, severe pre-eclampsia, (resting blood pressure ≥ 160mmHg systolic or 110 diastolic, recorded on at least two occasions 6 hours apart), known fetal anomaly, intrauterine infection, placental anomalies (previa, abruption, circumvallate, infarction), twins, and refusal of consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Uterine artery blood flow
Gestational age at delivery.

SECONDARY OUTCOMES:
Ductus venosus and MCA blood flow
Proprioceptive loss;
Maternal hemodynamic changes;
Fetal weight (throughout pregnancy and at delivery); amniotic fluid index;
obstetric outcome (maternal mortality, morbidity, neonatal mortality, morbidity, mode of delivery, obstetric complications).

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, BSc MBBS, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Hebrew University Medical Center, POB 12000, Jerusalem, Israel

REFERENCES:
- [Derived] Ginosar Y, Nadjari M, Hoffman A, Firman N, Davidson EM, Weiniger CF, Rosen L, Weissman C, Elchalal U; ACET study group. Antepartum continuous epidural ropivacaine therapy reduces uterine artery vascular resistance in pre-eclampsia: a randomized, dose-ranging, placebo-controlled study. Br J Anaesth. 2009 Mar;102(3):369-78. doi: 10.1093/bja/aen402. Epub 2009 Jan 27. PMID 19176534